CLINICAL TRIAL: NCT02310490
Title: A Controlled, Randomized, Within-subject, Multi-center Prospective Clinical Trial of DA-13-007 (Injectable Poly-L-lactic Acid) Versus SCULPTRA® Aesthetic (Injectable Poly-L-lactic Acid) in the Treatment of Nasolabial Fold Wrinkles.
Brief Title: DA-13-007 Versus Sculptra for the Treatment of Nasolabial Folds Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DermAvance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DermAvance DA-13-007
Record Dates: First submitted 2014-12-03; First posted 2014-12-08 (Estimated); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Face; Atrophy
Keywords: Nasolabial Folds
MeSH Terms: conditions — Facies; Atrophy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Right Side DA-13-007, Left Side Sculptra (Active Comparator): DA-13-007 right with left side Sculptra left side
  Interventions: Device: DA-13-007 right with left side Sculptra left side
- Left Side DA-13-007, Right Side Sculptra (Active Comparator): DA-13-007 left with Sculptra right side
  Interventions: Device: DA-13-007 left with left side Sculptra right side

INTERVENTIONS:
Device: DA-13-007 right with left side Sculptra left side — The treatment phase will consist of one to three visits at 3 week intervals during which eligible subjects will receive bilateral injections of study material in the left and right nasolabial fold wrinkles, including visits at weeks 3 and 6 for touch ups if needed
  Arms: Right Side DA-13-007, Left Side Sculptra
Device: DA-13-007 left with left side Sculptra right side — The treatment phase will consist of one to three visits at 3 week intervals during which eligible subjects will receive bilateral injections of study material in the left and right nasolabial fold wrinkles, including visits at weeks 3 and 6 for touch ups if needed
  Arms: Left Side DA-13-007, Right Side Sculptra

SUMMARY:
Study DA-13-007 is a randomized, evaluator-blinded, within subject (split face) multicenter clinical study of DA-13-007l (Injectable poly-l-lactic acid) compared to SCULPTRA in the treatment of nasolabial fold wrinkles. Qualifying subjects will be randomized to receive DA-13-007l and SCULPTRA on either the right or left side of the face.

DETAILED DESCRIPTION:
A randomized, evaluator-blinded, within subject (split face) multicenter clinical study of DA-13-007 (Injectable poly-l-lactic acid) compared to SCULPTRA in the treatment of nasolabial fold wrinkles. Qualifying subjects will be randomized to receive DA-13-007 and SCULPTRA on either the right or left side of the face. The treatment phase will consist of one to three visits at 3 week intervals during which eligible subjects will receive bilateral injections of study material in the left and right nasolabial fold wrinkles, including visits at weeks 3 and 6 for touch ups if needed. The follow-up phase will consist of assessments at 1, 3, 6, and 12 months after the last treatment, and safety and efficacy evaluations for an additional 12 months. Standardized photographs will be taken at screening and at all treatment phase and follow-up visits. Efficacy evaluations will be made by an on-site blinded evaluator, and of the photographs using a validated, standardized photo-numeric scale. The primary efficacy comparison between study treatments will be made on the mean change from baseline in the Wrinkle Severity Rating Scale of the nasolabial folds (as determined by the on-site blinded evaluator) and at the 12 month time point. Study participants will continue to be followed for safety and efficacy at months 18 and 24 after their last injection session.

ELIGIBILITY:
Inclusion Criteria:

* 1. Outpatient, male or female subjects of any race 21 years or older. Female subjects of childbearing potential must have a negative urine pregnancy test result at the Baseline Visit (test must have a sensitivity of at least 50U/mL for human chorionic gonadotropin) and practice a reliable method of contraception throughout the study.

  1. A female is considered of childbearing potential unless she is

     * postmenopausal for at least 12 months prior to study drug administration;
     * without a uterus and/or both ovaries; or
     * has been surgically sterile for at least 6 months prior to study drug administration.
  2. Reliable methods of contraception are:

     * hormonal methods or intrauterine device in use >30 days prior to study drug administration; or
     * barrier methods plus spermicide in use at least 14 days prior to study drug administration
     * vasectomized partner at least 3 months post operative or a zero sperm count post operatively 2. Demonstrate clinical evidence of moderate to severe bilateral aging in the nasolabial area, with wrinkles classified as a grade 3 or grade 4 on a 5-grade WSRS.

       3. Committed to abstain from procedures interfering with the treatment outcome (exclusion criteria) throughout the study.

       4. Able to understand the requirements of the study and sign Informed Consent and Photography Release forms.

Exclusion Criteria:

1. Pregnant (positive urine pregnancy test), are planning to become pregnant during the study period, have an infant they are breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
2. Subjects planning a facial cosmetic procedure during the study period or with prior cosmetic procedures (i.e., surgery) or visible scars that may affect the evaluation of response and/or quality of photography.
3. Facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, thick sebaceous skin, or an inability to substantially lessen upper facial rhytids even by physically spreading them apart.
4. Active skin disease within the treatment area within 6 months prior to study entry.
5. History of malignancy, excluding non-melanoma skin cancer within the past 5 years.
6. Profound atrophy/excessive weakness of muscles in target areas of injection.
7. History of facial nerve palsy.
8. Facial wrinkles therapy, such a permanent or enduring dermal fillers in the previous 2 years or bioresorbable during the previous 12 months.
9. Allergy or sensitivity to any component of the study medication (Section 8.1), or a known sensitivity to local anesthetics.
10. Previous botulinum toxin therapy within six (6) months of the Baseline Visit.
11. Use of systemic prednisone, penicillamine, anti metabolites or other bioequivalent collagen production inhibitors within 3 months of the Baseline Visit.
12. Has received (or is planning to receive) anti-coagulation, anti-platelet, or thrombolytic medications (e.g., warfarin), anti-inflammatory drugs (oral/injectable corticosteroids or non-steroidal anti inflammatory, eg.,aspirin, ibuprofen), or other substances known to increase coagulation time (e.g., Vitamin E, garlic, gingko). To clarify, no non-steroidal anti inflammatory e.g. asprin or ibuprofen within 10 days prior to injections or 3 days post injection.
13. Evidence of recent alcohol or drug abuse.
14. Medical and/or psychiatric problems that, in the Investigator's opinion, is severe enough to interfere with the study results.
15. History of poor cooperation, non-compliance with medical treatment, or unreliability.
16. Participation in an investigational drug or investigational device study within 3 months of the Baseline Visit.
17. A history of connective tissue disease (rheumatoid Arthritis, arthritis, lupus).
18. A history of multiple severe allergies or a history of anaphylactic shock.
19. Patients with a known history of or susceptibility to keloid formation or hypertrophic scarring.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Efficacy of treatment vs Comparator (using a 5-grade WSRS (wrinkle severity rating scale) score and a rating by an independent evaluator) | One Year
  To evaluate the efficacy of treatment versus the comparator in a non-inferiority statistical model using a 5-grade WSRS (wrinkle severity rating scale) score and a rating by an independent evaluator

SECONDARY OUTCOMES:
To evaluate the Global aesthetic improvement as assessed by investigators and subjects | Two Year
  • To evaluate the Global aesthetic improvement (GAI) as assessed by investigators and subjects
To evaluate subjects satisfaction using a six point subject satisfaction questionnaire. | Two Year
  To evaluate subjects satisfaction using a six point subject satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: William Werschler, MD, Principal Investigator — Premier Clinical Research
Locations (4):
- United States (4):
  - Bay Area Dermatology, Bradenton, Florida
  - Miami Skin Institute, Coral Gables, Florida
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - PCR, Spokane, Washington